CLINICAL TRIAL: NCT01132898
Title: Long Term Clinical Correlates of TBI: Imaging, Biomarkers, and Clinical Phenotyping Parameters
Brief Title: Long-term Clinical Correlates of Traumatic Brain Injury
Status: Terminated | Type: Observational
Why Stopped: At the discretion of the IRB
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 100118; 10-CC-0118
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Biomarkers; Functional Level; DTI; Neuropsychological Assessment; Natural History
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- cross-sectional TBI: Participants with a mild, moderate, or severe Traumatic Brain Injury enrolled within 5 years from injury. Seen at only one visit.
- HV: Healthy Volunteer with no history of TBI
- Prospective TBI: Participants with a mild, moderate, or severe Traumatic Brain Injury enrolled within 1 year from injury.
- Remote Select Exposure Samples: Participants who are unable to travel to the NIH Clinical Center to participate can remote consent, answer questionnaires remotely, and have biospecimens sent to our lab for analysis.
- Select Exposure Group: US government associated personnel experiencing TBI-like symptoms arising after possible exposure to a non-natural energy source
- Select Exposure Matched Unaffected: a longitudinal control group comprised of unaffected volunteers matched to the Select Exposure group

SUMMARY:
Background:

- Traumatic brain injury may have a range of effects, from severe and permanent disability to more subtle functional and cognitive deficits that often go undetected during initial treatment. To improve treatments and therapies and to provide a uniform quality of care, researchers are interested in developing more standardized criteria for diagnosing and classifying different types of traumatic brain injury. By identifying imaging and other indicators immediately after the injury and during the initial treatment phrase, researchers hope to better understand the nature and effects of acute traumatic brain injury.

Objectives:

- To study the natural history of traumatic brain injury by examining the changes in brain scans, blood samples, and brain function over 5 years after injury.

Eligibility:

- Individuals 18 years of age and older who have had a traumatic brain injury within the past 1 year.

Design:

* This study will include about eight visits to the NIH Clinical Center over 5 years. Participants will have four visits in the first year, and one visit each year for the following 4 years. Each visit will take between 1 and 4 days, and participants will be in the outpatient clinic for about 8 hours each day of the visit.
* At each study visit, participants will have some or all of the following tests:
* Medical history and physical examination
* Blood and urine tests
* Questionnaires and assessments of thinking and memory, which may be spoken aloud, written down, or entered into a computer
* Imaging scans, such as magnetic resonance imaging (MRI) or positron emission tomography/computed tomography (PET/CT).
* This study does not provide treatment and does not replace any current therapies. However, participants who are eligible for other National Institutes of Health studies may be referred to these studies by researchers.

DETAILED DESCRIPTION:
Objective

The primary objective is to contribute to the understanding of non-penetrating traumatic brain injury (TBI) through the description of the relationships between neuroimaging, hematological, and extensive functional/cognitive phenotyping measures. We will generate natural history data for cohort-based comparisons and to serve as the basis for future hypothesis-driven protocols. In addition, we will create and test a series of new taxonomies to describe TBI severity and predict outcome.

Study Population

Three hundred adult subjects with a clinical diagnosis of non-penetrating TBI (mild, moderate and severe) will be enrolled. Subjects will be recruited from NIH, affiliated hospitals/clinics, and in the community. One hundred adult healthy volunteers without a history of TBI will be seen for comparison. Additionally, a select group of up to 115 US government associated personnel experiencing TBI-like symptoms arising after possible exposure to a non-natural energy source, will be studied (select exposure group). This select group will require a separate age and sex matched group of 115 unaffected volunteers. Participants (100) who are not able to travel to the NIH Clinical Center to participate in the Select Exposure Group study can complete study tests and questionnaires remotely, and have biospecimens sent to our lab for analysis, as part of the remote select exposure samples group.

Design

This is a natural history study following a prospective cohort of subjects with a clinical diagnosis of non-penetrating traumatic brain injury with a cross-sectional sub-study. Subjects will be enrolled in the prospective cohort within one year of their head injury and then followed periodically for five years, with neuroimaging, including Magnetic Resonance Imaging (MRI), hematological, and extensive functional/cognitive phenotyping measures. Subjects will be enrolled in the cross-sectional sub-study within five years of their head injury and may be evaluated with MRI, hematological, and functional/cognitive measures usually within a single visit. However, procedures may be scheduled during multiple visits, depending on the number of procedures performed. Study participants may be offered standard of care rehabilitation therapies provided at no cost by Investigators and supervised by Dr. Chan. Tests will be subject to investigator discretion and subject willingness to participate in evaluation. After first MRI, future MRIs will be obtained based on subject willingness and investigator discretion from findings on previous imaging. Subjects will be stratified according to findings into cohorts for comparison. Subjects will not be treated with experimental therapies as part of the research study. This study will provide direct benefit to subjects as they will receive sensitive neuro-imaging and clinical testing that may have diagnostic value and rehabilitation therapies that might not be provided to them in the community. In addition to the TBI patient group, a longitudinal control group comprised of healthy volunteers will be collected. The control group participants may complete the Neuroimaging (MRI without gadolinium), hematological and functional/cognitive phenotyping measures as the TBI patient population.

The prospective select exposure group of US government associated personnel will be followed periodically for a total of six years. Subjects may complete neuroimaging, including Magnetic Resonance Imaging (MRI), hematological, and extensive functional/cognitive, auditory, vestibular, and oculomotor phenotyping measures. In addition to the select exposure group, a longitudinal control group comprised of unaffected volunteers matched to this group will be collected. The control group participants will complete the same Neuroimaging (MRI without gadolinium), hematological and functional/cognitive phenotyping measures as the select exposure patient population. Additionally, if a select exposure matched control participant is subsequently exposed, they may enroll into the select exposure group arm of the study for pre and post exposure analysis. Participants who are unable to travel to the NIH Clinical Center to participate can remote consent, answer questionnaires remotely via telephone or electronic communication methods, and have biospecimens sent to our lab for analysis. Participants enrolled in the any arm of the study who are unable to travel to NIH for any study visit may be asked to answer questions electronically (telephone, email, videoconferencing if within the US, etc) to allow for some data collection to occur at each time point.

Outcome Measures

A variety of outcome measures may be used including MRI, to include Diffusion Tensor Imaging (DTI), Dynamic Susceptibility Contrast (DSC), and functional Magnetic Resonance Imaging (fMRI), high field 7T MRI. In addition, extensive and sensitive clinical phenotyping will be performed to assess functional and cognitive impairment, including auditory, vestibular, and oculomotor testing, and quality of life assessments. Blood and saliva (buccal cells may be collected in lieu of whole blood for subjects unwilling or unable to provide blood draw) may also be collected and sent to a biorepository for future analysis if subject agrees to participation in sample collection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects eligible for participation in the TBI prospective cohort must meet the following inclusion criteria:

* Diagnosis of non-penetrating mild, moderate, or severe TBI
* Injury occurred less than one year before enrollment
* Age 18 years of age and older
* Able to provide informed consent or with a legally-authorized representative able to provide consent

Subjects eligible for participation in the cross-sectional sub-study must meet the following inclusion criteria:

* Diagnosis of non-penetrating mild, moderate, or severe TBI
* Injury occurred less than five years before enrollment
* Age 18 years of age and older
* Able to provide informed consent or with a legally-authorized representative able to provide consent

Subjects eligible for participation in the healthy volunteer control group must meet the following inclusion criteria:

* Age 18 and older
* Able to provide written informed consent
* Able to lie flat for up to 2 hours
* Good general medical and psychological health based on History and Physical (H&P)

Subjects eligible for participation in the Select Exposure prospective cohort must meet the following inclusion criteria:

* Referral from US State Department, Department of Health and Human Services or other governmental entity based on their assessment of symptomatology and potential exposure (may include, for example, abnormal auditory sensations and subsequent oculomotor, vestibular, and cognitive symptoms)
* Age 18 years of age and older
* Able to provide informed consent or with a legally-authorized representative able to provide consent

Subjects eligible for participation in the Select Exposure Matched Unaffected volunteer control group must meet the following inclusion criteria:

* Age 18 and older
* Able to provide written informed consent
* Good general medical and psychological health based on History and Physical (H&P)

Subjects eligible for participation in the Remote Select Exposure Samples cohort must meet the following inclusion criteria:

* Referral from US State Department, Department of Health and Human Services or other governmental entity based on their assessment of symptomatology and potential exposure (may include, for example, abnormal auditory sensations and subsequent oculomotor, vestibular, and cognitive symptoms)
* Age 18 years of age and older
* Able to provide informed consent (telephone or electronic signature)

EXCLUSION CRITERIA:

Subjects are not eligible for participation in the prospective cohort if any of the following conditions exist:

* Contraindication to MRI scanning including certain metal implants or devices such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitroglycerine) that cannot be removed for the study, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal imbedded in a patient s body (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near the patient s eyes).
* Multiple trauma or accidents in the past with non-certainty that metal objects are still present in the body
* Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
* Pregnant women.
* Women who are breast-feeding may enroll in the study, but will not receive PET-MRI.
* Inability to read or speak enough English to complete the clinical phenotyping testing.
* Medical or Psychological instability such that the subject could not reasonably be expected to fulfill the study requirements.
* Penetrating head injury.

Subjects are not eligible for participation in the cross-sectional sub-study if any of the following conditions exist:

* Contraindication to MRI scanning including certain metal implants or devices such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitroglycerine) that cannot be removed for the study, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal imbedded in a patient s body (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near the patient s eyes).
* Multiple trauma or accidents in the past with non-certainty that metal objects are still present in the body
* Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
* Pregnant women.
* Inability to read or speak enough English to complete the clinical phenotyping testing.
* Medical or Psychological instability such that the subject could not reasonably be expected to fulfill the study requirements.
* Penetrating head injury.

Subjects are not eligible to participate in the Select Exposure cohort if any of the following conditions exist:

* Pregnant women, may enroll in the study, but will not receive an MRI.
* Women who are breast-feeding may enroll in the study, but will not receive contrast MRI (gadolinium).
* Inability to read or speak enough English to complete the clinical phenotyping testing
* Medical or Psychological instability such that the subject could not reasonably be expected to fulfill the study requirements (such schizophrenia, uncontrolled hypertension, serious heart, lung, or kidney disease, or other condiditon that would make participation unsafe)

Subjects are not eligible for participation in the healthy volunteer control group if any of the following conditions exist:

* Contraindication to MRI scanning including certain metal implants or devices such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitroglycerine) that cannot be removed for the study, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal imbedded in a patient s body (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near the patient s eyes).
* Pregnant women
* Inability to read or speak enough English to complete the clinical phenotyping testing.
* History of a head injury, regardless of cause:.(Causes including: vehicle/bicycle accidents, falls, sports injuries, firearm injuries, blast injuries, violent shaking, etc)
* Weight more than 250 lbs.
* Height greater than 6 4
* Any current or prior alcohol or substance abuse.

Heavy alcohol use: The Substance Abuse and Mental Health Services Administration (SAMHSA) defines heavy alcohol use as binge drinking on 5 or more days in the past month. SAMHSA defines binge drinking as 5 or more alcoholic drinks for males or 4 or more alcoholic drinks for females on the same occasion (i.e., at the same time or within a couple of hours of each other) on at least 1 day in the past month.

Subjects are not eligible for participation in the Select Exposure Matched Unaffected volunteer group if any of the following conditions exist:

* Pregnant women, may enroll into the study but will not receive an MRI
* Inability to read or speak enough English to complete the clinical phenotyping testing.
* Any current or prior heavy alcohol or substance use.
* Have a medical or psychological condition, such schizophrenia, uncontrolled hypertension, serious heart, lung, or kidney disease, or other condition that would make it difficult for to do the study tests, might make participation unsafe, or would interfere with the study result

Subjects are not eligible for participation in the Remote Select Exposure Samples group if any of the following conditions exist:

* Have a blood disorder (such as anemia, bleeding disorders such as hemophilia, blood clots, and blood cancers such as leukemia, lymphoma, and myeloma) which would make participation in a blood draw dangerous, or would interfere with the study results
* Have a medical or psychological condition, such schizophrenia, uncontrolled hypertension serious heart, lung, or kidney disease, or other condition that would make it difficult to complete the study tests, might make participation unsafe, or would interfere with the study result

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three hundred adult subjects with a clinical diagnosis of non-penetration TBI will be enrolled. One hundred healthy volunteers without a history of TBI will be recruited to compare outcomes to TBI participants. A select exposure group of up to 115 US government associated personnel experiencing TBI-like symptoms arising after possible exposure to a non-natural energy source will be studied. An age and sex matched cohort of non TBI healthy volunteers will be recruited for comparison (n=115). One hundred participants who are unable to travel to the NIH Clinical Center to participate but would like to participate in the study can answer questionnaires remotely, and have biospecimens sent to our lab for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be to observe changes in the TBI Common Data Elements over time. | 30, 90, 180 days post injury, then annually out to 5 years.
  See NINDS Common Data Elements for TBI

SECONDARY OUTCOMES:
Changes in other clinical phenotyping measures over time | 30, 90, 180 days post injury, then annually out to 5 years.
  Comprehensive clinical phenotyping assessments

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CC-0118.html